CLINICAL TRIAL: NCT06387446
Title: Allogeneic Valve Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sitaram Emani, Associate Professor of Surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-P00044611
Record Dates: First submitted 2023-06-21; First posted 2024-04-29 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Valve Heart Disease; Valve Disease, Heart; Valve Disease, Aortic
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valve transplantation group (Experimental): This arm undergoes Allogeneic Valve transplantation
  Interventions: Procedure: Valve transplant

INTERVENTIONS:
Procedure: Valve transplant — Heart valves from an organ donor will be transplanted into recipient

SUMMARY:
Valves will be taken from hearts donated by organ donors, and implanted into patients who need a new heart valve.

DETAILED DESCRIPTION:
Heart valves in children and young adults may need replacement or repair. In many children the options for heart valve replacement do not grow as the child grows. A transplanted valve may have the option to grow with time and may reduce the need for multiple operations over a lifetime. This trial will study the outcomes of heartfelt transplant in children and young adults undergoing this procedure. The study will look at outcomes of valve transplant and any potential side effects.

ELIGIBILITY:
Inclusion Criteria

* Patients requiring aortic, pulmonary, mitral or tricuspid valve replacement.
* Pediatric patients 30 days or older and < 18 years, and adult patients 18-50 yrs.

  o Particularly patients with significant growth potential
* Insufficient options are available for valve replacement

  o Patients at risk of immunogenic bio-prosthetic valve failure
* Discussion with patient /family - option for durable valve rather than traditional prosthesis
* ABO compatible
* Patient and family able to travel to BCH within 48 hour time frame or within our organ procurement organization
* Patients that are able to maintain follow-up at BCH during the duration of the study
* Patients that are able to provide medical record authorization for 5 year follow-up

Exclusion Criteria

* Age < 30 days
* Irreversible multisystem organ failure; or additive effects of the multiple systems affected making transplant survival unlikely
* Progressive systemic disease with early mortality (genetic/metabolic, idiopathic, syndromic)
* Morbid obesity (BMI>35)
* Diabetes mellitus with evidence of end-organ damage
* Severe chromosomal, neurologic or syndromic abnormalities
* Immunocompromised condition (DiGeorge, SCID etc.)
* Active infection
* History of endocarditis
* HIV or chronic hepatitis B or C infection
* Malignancy within 5 years prior to transplant
* Severe renal or liver failure
* Inadequate social support for post-transplant management
* Recent history of illicit drug, tobacco or alcohol abuse despite trials/assistance to stop behavior
* Evidence of large stroke with high risk for hemorrhagic conversion
* Heart transplant recipient
* Patients that are unable to follow-up during the initial 6 month window
* Patients that are unable to provide medical record authorization for 5 years

Ages: 30 Days to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Valve Regurgitation | One year
  Heart valve regurgitation by echocardiogram. The degree of regurgitation is read and quantified by an echocardiologist.
Valve Annulus Growth | One Year
  Measurement of valve annulus via echocardiogram, CT scan and MRI. This will be quantified by whether or not the annulus continues to increase in size as the subject grows.
Leaflet Growth | One Year
  Measurement of leaflet height via echocardiogram, CT scan and MRI and reviewed by an echocardiologist. This will be analyzed by whether or not the leaflets continue to grow in size, with the subject.

SECONDARY OUTCOMES:
Ventricular Function | One year
  Ventricular function will be visualized using echocardiogram, measured as ejection fraction as well as shortening fraction and will be determined by an echocardiologist. The factors involved will be the symmetrical squeeze of the ventricles, the ejection fraction, ventricular end systolic and diastolic volume with calculation of stroke volume to come to a surrogate of cardiac output.
Survival | 5 years
  The number of patients that survive the initial procedure and long term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sitaram Emani, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No